CLINICAL TRIAL: NCT03390361
Title: Intraindividual Comparison of Proinflammatory Cytokines (IL-1β, IL-6) and Total-prostaglandin (PG) Following Femtosecond Laser-assisted Cataract Surgery Using a Low-energy, High-frequency Femtosecond Laser-Device Compared to Manual Cataract Surgery
Brief Title: Release of Proinflammatory Cytokines (IL-1β, IL-6) and Total-prostaglandin (PG) Following Femtosecond Laser-assisted Cataract Surgery Compared to Manual Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Clinical Professor, Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Femto IL + PG Study
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Age Related Cataracts
Keywords: Laser Cataract Surgery; Prostaglandin

STUDY DESIGN:
Intervention Model Description: Patients' eyes will be randomized into two groups receiving either MCS or LCS. In the LCS group aqueous humour will be collected exactly five minutes after laser pretreatment. In the MCS group aqueous humour will be collected before manual manipulation of anterior chamber. Aqueous humour will be screened with Enzyme-linked Immunosorbent Assay (ELISA) Kits for Interleukin-1β; Interleukin-6 and PG.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Groups will be randomized. Randomization information will be put in a sealed envelope on screening date and opened in operating theatre right before the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCS (Active Comparator): Laser cataract surgery will be performed. 5-minutes after LCS aqueous humour will be collected and frozen in -80° celsius.
  Interventions: Device: Femtosecond Laser-assisted
- MCS (Placebo Comparator): Manual cataract surgery will be performed. Aqueous humour will be collected and frozen in -80° celsius before MCS starts.
  Interventions: Procedure: Manual Cataract Surgery

INTERVENTIONS:
Device: Femtosecond Laser-assisted — Laser cataract surgery will be performed in one eye
  Arms: LCS
Procedure: Manual Cataract Surgery — Manual cataract surgery will be performed in contralateral eye
  Arms: MCS

SUMMARY:
Patients with bilateral age related cataract will be included in the study. Manual cataract surgery (MCS) will be performed in one eye and laser cataract surgery (LCS) in the corresponding eye. LCS will be performed with an approved femtosecond laser (FSL) device with an integrated imaging system.

After surgery aqueous humour will be collected and screened with Enzyme-linked Immunosorbent Assay (ELISA) Kits for Interleukin-1β; Interleukin-6 and PG.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract necessitating phacoemulsification extraction and posterior intraocular lens implantation.
* Pupil dilation of ≥ 6.5mm
* Age 40 and older

Exclusion Criteria:

* Corneal abnormality
* Pseudoexfoliation
* Preceding ocular surgery or trauma
* Uncontrolled glaucoma
* Proliferative diabetic retinopathy
* Iris neovascularization
* History of uveitis/iritis
* Microphthalmus
* Recurrent intraocular inflammation of unknown etiology
* Blind fellow eye
* Uncontrolled systemic or ocular disease
* Pregnancy
* Lactation

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2016-08-09 (Actual); Study Completion 2016-11-25 (Actual)

PRIMARY OUTCOMES:
Proinflammatory cytokines (IL-1β, IL-6) and total-PG | 5 minutes after laser procedure
  Interleukin IL-1β, Interleukin IL-6, total-prostaglandin

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Menapace, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No